CLINICAL TRIAL: NCT05603039
Title: A Phase Ib/II Trial to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of QL1706 or QL1604 Combined With Bevacizumab in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Phase Ib/II Trial to Evaluate the Safety and Efficacy of QL1706 in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-106
Record Dates: First submitted 2022-10-21; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Advanced Liver Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QL1706(5mg/kg) (Experimental): QL1706(5mg/kg) Combined with Bevacizumab
  Interventions: Drug: QL1706; Drug: Bevacizumab
- QL1604 (Experimental): QL1604 Combined with Bevacizumab
  Interventions: Drug: QL1604; Drug: Bevacizumab
- QL1706(7.5mg/kg) (Experimental): QL1706(7.5mg/kg) Combined with Bevacizumab
  Interventions: Drug: QL1706; Drug: Bevacizumab

INTERVENTIONS:
Drug: QL1706 — 5 mg/kg#D1#Q3W IV or 7.5 mg/kg#D1#Q3W IV
  Arms: QL1706(5mg/kg); QL1706(7.5mg/kg)
Drug: QL1604 — 200mg#D1#Q3W IV
  Arms: QL1604
Drug: Bevacizumab — 15 mg/kg#D1#Q3W IV or 7.5 mg/kg#D1#Q3W IV

SUMMARY:
This is a phase Ib/II trial to evaluate the safety, pharmacokinetics and preliminary efficacy of QL1706 or QL1604 combined with bevacizumab in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is an open, multicenter phase Ib/II trial of QL1706 or QL1604 combined with bevacizumabin patients with advanced hepatocellular carcinoma to evaluate the safety, PK characteristics and preliminary efficacy. This trial is divided into three cohorts, Cohort A, Cohort B and Cohort C.

Cohort A was the dose exploration phase of the study, with 2 dose groups designed, QL1706 5mg/kg q3w + bevacizumab 7.5mg/kg q3w group and QL1706 5mg/kg q3w + bevacizumab 15mg/kg q3w group, to explore the safe dose of bevacizumab.

After approximately 20 cases are enrolled in the bevacizumab safety dose group identified in Cohort A, enrollment will be initiated in Cohort B. Cohort B will be QL1604 200 mg fixed dose q3w + bevacizumab safety dose, and random enrollment will be used for both Cohort A and Cohort B.

The decision to initiate a cohort C study will be based on the preliminary results of the efficacy analysis of cohort A and cohort B. If a Cohort C study is initiated, the Cohort C dosing regimen will be QL1706 7.5 mg/kg q3w + bevacizumab safe dose q3w.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participated voluntarily and signed an informed consent form.
2. Age ≥ 18 years old at the time of signing the informed consent form, male or female.
3. Advanced hepatocellular carcinoma diagnosed by histopathology or clinical diagnosis, with disease unsuitable for radical surgery and/or local treatment, or disease progression after surgery and/or local treatment.
4. No prior systemic treatment for HCC.
5. Child-Pugh liver function classification of grade A versus better grade B.
6. Eastern Cooperative Oncology Group (ECOG) physical status score of 0-1.
7. Expected survival ≥ 3 months.

(9) Functional level of vital organs must be compliant prior to first administration of trial drug.

(10) Subject agrees to use effective contraception for contraception from the time of signing the informed consent until 180 days after the last use of the trial drug. Females of childbearing age cannot be in pregnancy or breastfeeding.

Exclusion Criteria:

1. Subjects with symptomatic CNS metastases were not allowed to be enrolled.
2. Patients with a history of other malignancies within 5 years prior to signing informed consent.
3. Active autoimmune disease that may have worsened during the course of receiving study drug therapy.
4. Concomitant disease that interferes with the subject's ability to complete the study.
5. History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
6. HIV-positive patients; HCV antibody-positive and HCV RNA-positive patients; patients with co-infection with HBV and HCV.
7. Patients with a known history of psychotropic substance abuse, alcoholism, or drug use
8. Those who have participated in other clinical studies and have used other clinical trial drugs within 4 weeks prior to the use of the trial drug
9. Prior immunotherapy or prior targeted therapy.
10. PCP treatment requires 2 weeks of elution before enrollment and is prohibited during the trial.
11. Known previous hypersensitivity to macromolecular protein agents, or any component of the test drug.
12. Live vaccination within 4 weeks prior to the first administration of the test drug.
13. History of hemoptysis, or history of gastrointestinal bleeding, intestinal obstruction and/or previous clinical signs or symptoms of gastrointestinal obstruction.
14. Abdominal or bronchoesophageal fistula, gastrointestinal perforation or intra-abdominal abscess, major vascular disease.
15. Current or recent treatment with aspirin, clopidogrel, or current or recent treatment with dipyridamole, ticlopidine, and cilostazol; use of anticoagulation therapy for therapeutic purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | up to 1year
  The ORR assessed according to RECIST v1.1

SECONDARY OUTCOMES:
Duration of remission (DOR) Duration of remission (DOR) Duration of remission (DOR) Duration of remission (DOR) | Every 6 weeks up to 48 weeks during study, and every 12 weeks after the end of treatment up to 1year.
  The DOR assessed according to RECIST v1.1

OTHER OUTCOMES:
Disease Control Rate (DCR) Disease Control Rate (DCR) Disease Control Rate (DCR) | Every 6 weeks up to 48 weeks during study, and every 12 weeks after the end of treatment up to 1year.
  The DCR assessed according to RECIST v1.1
Progression free survival (PFS) | Every 6 weeks up to 48 weeks during study, and every 12 weeks after the end of treatment up to 1year.
  The PFS and progression-free survival at 6 and 12 months (PFS6/12)
Overall survival (OS) | From date of randomization until the date of death from any cause, , 12 months after the last use of the trial drug, or study completion/closure, whichever came first.
  The Overall survival and 1-year OS rate Overall survival Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No